CLINICAL TRIAL: NCT06239935
Title: Early Rehospitalization of Persons Aged 75 Years or Older Admitted to a Geriatric Post-emergency Unit: Rates and Predictive Factors
Brief Title: Early Rehospitalization of Persons Aged 75 Years or Older Admitted to a Geriatric Post-emergency Unit.
Acronym: BACK-UPUG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 23_0359
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Early Rehospitalization of the Elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The older population is increasing, and one of the challenges is to prevent functional disability. Longer hospital stays are a recognized factor in dependency. Older subjects may present multiple complications, and therefore be frequently readmitted to hospital. Readmission to hospital is a costly and iatrogenic event in terms of independence, and must therefore be limited. The most vulnerable older patients therefore require specific care to avoid these iatrogenic complications, and various innovative structures have been developed, such as mobile geriatric teams, carrying out assessments in emergency departments, or geriatric post-emergency units with a shorter length of stay to reduce the iatrogenic impact of hospitalization.In November 2022, a temporary hospitalisation unit based on this model was opened at the CHU d'Angers with 11 beds. The aim of this study is to estimate the rate of early rehospitalisation (< 30 days) between December 2022 and September 2023, and the factors associated with it. Once identified, these factors will allow us to further select patient profiles that are suitable for care in these very short stay units.

ELIGIBILITY:
Inclusion Criteria:

- Patient admitted to the temporary geriatric hospitalization unit between December 1, 2022 and September 30, 2023

Exclusion Criteria:

* Patients moved to another medical, surgical or obstetrics department of the Angers University Hospital during their stay.
* Death during stay.
* Patient assigned to a unit other than the temporary geriatric hospitalization unit.
* Patient already hospitalized in the unit during the recruitment campaign.
* Opposition to data use

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the geriatric post-emergency medicine unit at angers university hospital
Sampling Method: Non-Probability Sample
Enrollment: 687 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Early rehospitalization (< 30 days after hospital discharge) | 30 days
  Early rehospitalization (< 30 days after hospital discharge)